CLINICAL TRIAL: NCT03313336
Title: A Double-blind, Randomized, 2-period, Placebo-controlled, Single-center, Crossover Study to Assess the Therapeutic Equivalence of the EMLA Current Reference Patch and the EMLA Test Patch in Healthy Subjects.
Brief Title: A Study to Assess Therapeutic Equivalence Between Test EMLA Patch With Marketed EMLA Patch in Healthy Subjects.
Acronym: EMLA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: D069GC00001
Record Dates: First submitted 2017-09-08; First posted 2017-10-18 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Pain
Keywords: Dermal anesthesia.; Venipuncture and intravenous cannulation.; Skin blanching or erythema.; Phase I.; Therapeutic equivalence.; Eutectic Mixture of Local anaesthetics (EMLA)
MeSH Terms: conditions — Pain; Erythema

STUDY DESIGN:
Intervention Model Description: This study will be a double-blind, randomized, 2-period, placebo-controlled, crossover study in healthy male and female subjects, performed at a single study center. Prior to inclusion, informed consent will be obtained. A brief medical history, including limited demographic data (gender, age and ethnicity) will be recorded, and eligibility for inclusion to the study will be established through a physical inspection of hands. Subjects will be shown how to complete the visual analogue scale (VAS). At each specific study visit, each subject will undergo a left-right comparison of two patch preparations, followed by a repeated test with an alternate combination of preparations. Thus, the study will comprise: Visit 1: EMLA Test Patch plus Placebo Patch OR EMLA Test Patch plus EMLA current Reference Patch. Visit 2: EMLA Test Patch plus EMLA current Reference Patch OR EMLA Test Patch plus Placebo Patch.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): EMLA Test Patch.
  Interventions: Drug: EMLA test patch
- Cohort 2 (Active Comparator): EMLA Reference Patch.
  Interventions: Drug: EMLA current reference patch
- Cohort 3 (Placebo Comparator): Placebo patch.
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: EMLA test patch — EMLA® Test Patch containing the active ingredients lidocaine base 25 mg/g and prilocaine base 25 mg/g in an oil-in-water emulsion saturating the absorbent cellulose disc. The source of cellulose for the cellulose disc will be provided from a new supplier in this test patch.
  Arms: Cohort 1
Drug: EMLA current reference patch — EMLA current Reference Patch, containing the active ingredients lidocaine base 25 mg/g and prilocaine base 25 mg/g in an oil-in-water emulsion saturating the absorbent cellulose disc.
  Arms: Cohort 2
Drug: Placebo Patch — Placebo Patch, based on the EMLA Test Patch (incorporating the absorbent cellulose disc with cellulose from the current supplier), where the absorbent disc will be saturated with a placebo oil-in-water emulsion, where the eutectic mixture of lidocaine and prilocaine is replaced with fractionated coconut oil and chlorhexidine digluconate 20%, with identical appearance to the active EMLA patches.
  Arms: Cohort 3

SUMMARY:
A double-blind, randomized, 2-period, placebo-controlled, single-center, crossover study, efficacy study demonstrating the therapeutic equivalence of the test cellulose disc (matrix) in EMLA patch and the current commercial cellulose disc (matrix) in EMLA patch in healthy subjects.

DETAILED DESCRIPTION:
This study will be a double-blind, randomized, 2-period, placebo-controlled, crossover study in healthy male and female subjects, performed at a single study center. Prior to inclusion, informed consent will be obtained. A brief medical history, including limited demographic data (gender, age and ethnicity) will be recorded, and eligibility for inclusion to the study will be established through a physical inspection of hands. Subjects will be shown how to complete the VAS. Visual analogue scale (VAS) as a research tool is frequently used for the assessment of pain severity and relief. VAS is easy to use and can be applied in a variety of settings; results are reproducible. VAS data are sensitive to treatment effects and can be analyzed using parametric statistical techniques. At each specific study visit, each subject will undergo a left-right comparison of two patch preparations, followed by a repeated test with an alternate combination of preparations. Thus, the study will comprise: Visit 1: EMLA Test Patch plus Placebo Patch OR EMLA Test Patch plus EMLA current Reference Patch. Visit 2: EMLA Test Patch plus EMLA current Reference Patch OR EMLA Test Patch plus Placebo Patch. There will be a washout period of at minimum of 4 calendar days between treatment periods (visits). No follow-up visit is needed. Any adverse event (AE) that is ongoing at the last visit will be followed up as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and female subjects aged 18 to 60 years.
3. Have healthy skin over hands, with no inflammation or open wounds.
4. Able to understand, read and speak the German language.
5. Easy accessible veins on the dorsum of both hands.

Exclusion Criteria:

1. Current significant active skin disease such as widespread eczema or active atopic dermatitis.
2. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI, to local anesthetics of the amide type or to any of the components of the EMLA emulsion (e.g., castor oil polyoxyl hydrogenated).
3. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI to chlorohexidine (preservative in the placebo patch emulsion).
4. Subjects who previously entered this study.
5. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
6. Judgement by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
7. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Comparison of anesthetic efficacy of EMLA Test Patch with the marketed EMLA patch (EMLA current Reference Patch) by pain reduction assessment. | At test procedure 1 and at test procedure 2 (which is after 4 days of washout period following test procedure 1).
  To compare the anesthetic efficacy in pain reduction after an intravenous needle insertion whether or not actual IV insertion was achieved will be evaluated by visual analogue scale (VAS). The degree of pain experienced will be assessed on a 100 mm horizontal, non-graded paper-based VAS, with the endpoints representing "no pain" (0 mm), to "the worst possible pain" (100 mm). The VAS scores will be listed by subject, treatment sequence (TP/TR and TR/TP, where T=test, R=reference and P=Placebo), treatment (T, R and P) and hand (left, right).

SECONDARY OUTCOMES:
Number of participants with Adverse events (AEs), skin sensation and reactions as variables of safety and tolerability. | From randomization until test procedure 2 or last study visit, whichever is later.
  AEs will be collected from the start of randomization throughout the treatment period up to and including the Follow-up Visit. Any AE that is ongoing at the last visit will be followed up as appropriate. Serious AEs will be recorded from the time of informed consent. Local skin sensations will be assessed by asking about injection site sensations (sensation experienced before removal of the patch), this will be rated on a four-point scale: none, mild, moderate or severe. Skin reactions will be performed after removal of the patch to inspect the area which has been in contact with the cream and the patch. Two separate assessments will be made - one for the skin in contact with the cream and one for the skin which had been in contact with the adhesive border.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med.Rainard Fuhr, Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No